CLINICAL TRIAL: NCT05692128
Title: Frequency and Severity of Thrombocytopenia in Neonatal Sepsis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ragab Mohamed Amin Ghandour, Principal investigator, Assiut University
Other Study IDs: Thrombocytopenia neonatal seps
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Neonatal Sepsis
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Hematological and chemistry tests — Laboratory tests

SUMMARY:
The aim of our study was to find the frequency of thrombocytopenia and its severity in neonates with sepsis

DETAILED DESCRIPTION:
Early-onset sepsis remains a common and serious problem for neonates, especially preterm infants. Group B streptococcus (GBS) is the most common etiologic agent, while Escherichia coli is the most common cause of mortality. Current efforts toward maternal intrapartum antimicrobial prophylaxis have significantly reduced the rates of GBS disease but have been associated with increased rates of Gram negative infections, especially among very-low-birth-weight infants .

The diagnosis of neonatal sepsis is based on a combination of clinical presentation, the use of nonspecific markers, including C-reactive protein, blood cultures, CBC , ESR. .Its miles assessed that sepsis develops in 20% of neonates, of which 1% die in the early days... Empirical treatment should be based on local patterns of antimicrobial resistance but typically consists of the use of ampicillin and gentamicin or ampicillin and cefotaxime if meningitis is suspected, until the etiologic agent has been identified. Current research is focused primarily on development of vaccines against GBS. It encompasses various systemic infections of the newborn such as septicemia, meningitis, pneumonia, pyogenic arthritis, osteomyelitis and urinary tract infections. Sepsis is the commonest cause of neonatal mortality; it is responsible for about 30-50% of the total neonatal deaths in developing countries. It is estimated that up to 20% of neonates develop sepsis and approximately 1% die of sepsis related causes. Sepsis related mortality is largely preventable with rational antimicrobial the rapid and aggressive supportive care .

. Based on the onset, sepsis is divided into three categories: early-onset sepsis (fewer than three days of age), late-onset sepsis (LOS) (at 3-28 days of age), and late late-onset sepsis (at 29-120 days of age). Among all three types, late-onset sepsis (LOS) is frequent, particularly in VLBW neonates. One of the early indicators for neonatal sepsis is thrombocytopenia . Thrombocytopenia is one of the most common hematological disorders at newborn age, affecting the majority of neonates admitted to the NICU . Neonates admitted to NICUs develop thrombocytopenia in 20%-35% of all admissions, and a hike in percentage is noted with a drop in gestational age . The majority of neonates present with mild to moderate thrombocytopenia. Sepsis in the newborn is one of the chief causes of thrombocytopenia in neonates, and it can become very severe and can increase the risk of bleeding within 24 hours after developing an infection . The exact mechanism of low platelets in neonatal sepsis is unknown, but it has been proposed that sepsis causes endothelial injury, which in turn triggers the reticuloendothelial system. Platelet consumption exceeds production and causes thrombocytopenia . Thrombocytopenia and neonatal sepsis associations have been highlighted by recognizing thrombocytopenia as the prominent key risk feature for sepsis-related fatalities in neonates . An observational study by Noreen et al. showed that the frequency of thrombocytopenia is higher in neonates admitted to the NICU for any reason . Neonatal sepsis must not be considered as a homogenous entity, as it spurns both the pathogenic and clinical variations among numerous causative microorganisms and clinical syndromes and features of septicemia. No local study has been done in the recent past that emphasizes the incidence of thrombocytopenia in neonatal sepsis. In this research, we will present the characteristics of thrombocytopenia related to sepsis in both gram-negative and gram-positive cells. This will be beneficial for early diagnosis and treatment, predicting morbidity and mortality.

The results of this study will provide us with local statistics on the magnitude of neonatal thrombocytopenia in sepsis, and this will provide a window for further research

ELIGIBILITY:
Inclusion criteria:

* All neonates less than 28 days old, of both genders, and positive blood culture were included.

Exclusion criteria:

* Those with a mother's history of ITP, SLE, or other autoimmune disorders on medication during pregnancy (sulfonamides, quinine, quinidine, thiazides, tolbutamide, vancomycin, hydralazine, and heparin) and neonates with a history of bleeding disorders in the family, trisomies, or Turner/Noonan's syndromes were excluded. All neonates less than 28 days old, of both genders were included.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All neonates admitted to NICU sufferd from neonatal sepsis and have thrombocytopenia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Find out frequency of cases admited to NICU with neonatal sepsis and have thrombocytopenia and document it's severity | Baseline
  Detect frequency and severity of thrombocytopenia in cases admitted in NICU with neonatal sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Amal A Soliman, Study Chair — Assiut University

REFERENCES:
- [Background] Simonsen KA, Anderson-Berry AL, Delair SF, Davies HD. Early-onset neonatal sepsis. Clin Microbiol Rev. 2014 Jan;27(1):21-47. doi: 10.1128/CMR.00031-13. PMID 24396135